CLINICAL TRIAL: NCT00341224
Title: Steppin' Up: Positive Youth Development Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999903261; 03-CH-N261
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-12-09

CONDITIONS: Mentoring
Keywords: Aggression; Violence; Adolescents; Randomized Trial; Behavioral Intervention
MeSH Terms: conditions — Aggression

INTERVENTIONS:
Behavioral: Group-mentoring intervention — Group mentoring used to teach social skills to middle school students

SUMMARY:
As an antidote to juvenile aggression and violence, which has increased in recent years, group mentoring offers a viable alternative to intensive one-on-one mentoring. However, no group-mentoring programs have been evaluated.

The purpose of this study is to assess the efficacy of a school-based, group-mentoring intervention designed to prevent aggressive and deviant behavior among early adolescents.

Study participants will be incoming 6th grade students from two inner-city Baltimore middle schools and their parents. Approximately 1,400 students and their parents are expected to participate. All 6th grade students in these schools are eligible for the study.

Weekly student group-mentoring sessions are the principal component of this study. These groups will be held during the school day and will be designed to increase social skills and encourage academic engagement, restraint, and problem-solving. A master's level professional will direct and conduct these intervention activities, which will employ the use of field trips, cooperative games, discussion of real-life situations, and role playing.

Students will also complete a 1-hour written survey each fall and spring from grades 6-8 about the program and about attitudes and behaviors related to school involvement and staying healthy and safe. Study staff will contact participants' teachers and review their past and current school records, including attendance, grades, and disciplinary information.

Parents may be asked to participate in group meetings and will complete in-person or telephone interviews (about 20 minutes each) about similar information over a 3-year period (6th grade to 8th grade).

DETAILED DESCRIPTION:
Group mentoring offers a potentially viable alternative to intensive one-on-one mentoring. However, no group mentoring programs have been evaluated. The purpose of this study is to assess the efficacy of a school-based, group-mentoring intervention designed to prevent aggressive and deviant behavior among early adolescents. Two successive cohorts of incoming 6th grade students from two inner-city Baltimore middle schools and their parents will be randomized to comparison group or intervention group consisting of weekly group-mentoring sessions for youth and persuasive communication and small-group media-development projects for parents.

ELIGIBILITY:
* INCLUSION CRITERIA:

The population of interest for the randomized trial is 6th-grade students and their parents in two participating Baltimore middle schools. Participating schools are urban, inner-city schools located in neighborhoods with low SES and high rates of unemployment and crime.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-07-23; Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

PRIMARY OUTCOMES:
Student fighting | Immediate poste test, 12-month follow-up

SECONDARY OUTCOMES:
Academic engagement | Immediate post test, 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bailey SL, Flewelling RL, Rosenbaum DP. Characteristics of students who bring weapons to school. J Adolesc Health. 1997 Apr;20(4):261-70. doi: 10.1016/S1054-139X(96)00283-2. PMID 9098729
- [Background] DuRant RH, Krowchuk DP, Kreiter S, Sinal SH, Woods CR. Weapon carrying on school property among middle school students. Arch Pediatr Adolesc Med. 1999 Jan;153(1):21-6. doi: 10.1001/archpedi.153.1.21. PMID 9894995
- [Background] Ellickson PL, McGuigan KA. Early predictors of adolescent violence. Am J Public Health. 2000 Apr;90(4):566-72. doi: 10.2105/ajph.90.4.566. PMID 10754971